CLINICAL TRIAL: NCT05981040
Title: A Phase 2, Proof-of-concept, Placebo Controlled, Randomized, Multi-centre, Double Blind Study of ZYIL1 to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ZYIL1 in Patients With Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZYIL1.23.003
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — ZYIL1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Active Comparator): ZYIL1 capsules 25 mg for oral administration + matching placebo of 50 mg ZYIL1 capsule
  Interventions: Drug: ZYIL1 capsules 25 mg and 50 mg Placebo
- Arm 2 (Active Comparator): ZYIL1 capsules 50 mg for oral administration + matching placebo of 25 mg ZYIL1 capsule
  Interventions: Drug: ZYIL1 capsules 50 mg and 25 mg Placebo
- Arm 3 (Active Comparator): ZYIL1 capsules 25 mg for oral administration + ZYIL1 capsules 50 mg for oral administration
  Interventions: Drug: ZYIL1 capsules 25 mg and ZYIL1 capsules 50 mg
- Arm 4 (Placebo Comparator): Matching placebo of 25 mg ZYIL1 capsule + Matching placebo of 50 mg ZYIL1 capsule
  Interventions: Drug: Matching placebo 25 mg and Matching placebo 50 mg

INTERVENTIONS:
Drug: ZYIL1 capsules 25 mg and 50 mg Placebo — ZYIL1 capsules 25 mg for oral administration + matching placebo of 50 mg ZYIL1 capsule
  Arms: Arm 1
Drug: ZYIL1 capsules 50 mg and 25 mg Placebo — ZYIL1 capsules 50 mg for oral administration + matching placebo of 25 mg ZYIL1 capsule
  Arms: Arm 2
Drug: ZYIL1 capsules 25 mg and ZYIL1 capsules 50 mg — ZYIL1 capsules 25 mg for oral administration + ZYIL1 capsules 50 mg for oral administration
  Arms: Arm 3
Drug: Matching placebo 25 mg and Matching placebo 50 mg — Matching placebo of 25 mg ZYIL1 capsule + Matching placebo of 50 mg ZYIL1 capsule
  Arms: Arm 4

SUMMARY:
ZYIL1 is expected to show benefit in patients with Amyotrophic Lateral Sclerosis (ALS). The present study aims to determine the safety, tolerability, pharmacokinetics, and pharmacodynamics of ZYIL1 when administered to subjects with ALS.

DETAILED DESCRIPTION:
This is a proof-of-concept, placebo controlled, randomized, multi-centre,double blind study designed to evaluate the efficacy, safety, tolerability, pharmacokinetics, and pharmacodynamics in patients with Amyotrophic Lateral Sclerosis following a twice daily oral administration of ZYIL1 or matching placebo to patients aged between 18 and 80 years (inclusive at screening).

Treatment duration will be twelve (12) weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or female patients aged between 18 and 80 years (inclusive at screening).
2. Diagnosis of probable or definite ALS, according to the revised version of the El Escorial World Federation of Neurology criteria. Refer Appendix III - El Escorial Criteria.
3. Time since onset of first symptom of ALS ≤9 months
4. Slow Vital Capacity (SVC) ≥ 50% of the predicted value
5. Be able to swallow the study capsules during study
6. Either not currently receiving riluzole or on a stable dose of riluzole for at least 4 weeks before the screening visit. Participants receiving riluzole are expected to remain on the same dose throughout the duration of the study
7. Either not currently receiving edaravone or on edaravone treatment. Participants receiving edaravone must have completed at least 1 cycle of treatment before the screening visit and are expected to continue with stable dose edaravone treatment throughout the duration of the study.
8. Female patients must be non-pregnant, non-lactating and women of child-bearing potential/ sexually active women, unless surgically sterile (at least 6 months prior to study drug administration) or postmenopausal* for at least 12 consecutive months, must agree to use adequate contraception (hormonal contraceptives [combined estrogen and progestogen oral contraceptive, patch, contraceptive vaginal ring, injectable progestogen, and implants] or contraceptive subdermal implant or percutaneous contraceptive patches or intrauterine device [IUD] or intrauterine system [IUS]; vasectomy and tubal ligation or barrier method of birth control; female condom with spermicide, cervical cap, diaphragm with spermicide, contraceptive sponge), absolute sexual abstinence, use of condom with spermicide by sexual partner or sterile [at least 6 months prior to study drug administration], during study and up to 32 days after the last dose of study drug.

   *Postmenopausal defined as 12 months of spontaneous amenorrhea with an appropriate clinical profile (e.g., age appropriate, >45 years, in the absence of hormone replacement therapy).
9. All male patients should avoid fathering a child by either true abstinence, hormonal or barrier method (e.g., male condom with diaphragm, male condom with cervical cap) or with their sexual partner the use of effective means of contraception throughout and till 92 days of administration of the last dose. They must not donate sperm for at least 92 days after the last dose of study drug.
10. Ability to provide written informed consent and to be compliant with the schedule of protocol assessments. In case of illiterate patients, thumb impression of the patients will be obtained along with the signature of the impartial witness or legally authorized representative (LAR) on the consent form prior to patient's participation in the trial.Date of ALS Symptom Onset. For the purposes of this study, the date of symptom onset will be defined as the date the subject first had symptoms of their disease, i.e., weakness. To be eligible for this study, the date of symptom onset must be no greater than exactly 9 months prior to the Screening Visit date.

Exclusion Criteria:

1. With significant cognitive impairment, psychiatric disease, other neurodegenerative disorder (e.g., Parkinson disease or AD), substance abuse other causes of neuromuscular weakness, or any other condition that would make the participants unsuitable for participating in the study or could interfere with assessment or completing the study in the opinion of the Investigator.
2. History of recent serious infection (e.g., pneumonia, septicemia) within 4 weeks of the screening visit; infection requiring hospitalization or treatment with IV antibiotics, antivirals, or antifungals within 4 weeks of screening; or chronic bacterial infection (such as tuberculosis) deemed unacceptable as per the Investigator's judgment
3. With active herpes zoster infection within 2 months prior to the screening visit
4. A documented history of attempted suicide within 6 months prior to the screening visit, or in the Investigator's judgment are at risk for a suicide attempt
5. History of unstable or severe cardiac, pulmonary, oncological, hepatic, or renal disease or another medically significant illness other than ALS precluding their safe participation in this study
6. Participants who are pregnant or are currently breastfeeding
7. A known history of allergy to any ingredients of ZYIL1
8. Patients taking concomitant medicines within 7 days or 5 half-lives of the medication (whichever is longer) prior to first dose of study drug administration till end of the study, which are substrate of CYP1A2 enzymes (e.g., alosetron, caffeine, duloxetine, melatonin, ramelteon, tasimelteon, tizanidine etc.) and CYP2B6 enzymes (e.g., bupropion, efavirenz etc.).
9. Use of any steroids, colchicine or anti-IL-1 inhibitors within 7 days or 5 half-lives of the medication (whichever is longer) prior to first dose of study drug administration.
10. Use of any investigational drugs concurrently or within 4 weeks or 5 half-lives (whichever is longer), prior to first dose of study drug administration.
11. Any clinically significant and/or laboratory significant value or other instability that would prevent the patient from participating in the study as determined by the Investigator.
12. Received a live vaccine within 14 days before the screening visit or planning to receive during the study
13. Participants who have received stem cell or gene therapy for ALS at any time in the past
14. Any of the following laboratory values at screening

    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3.0 × upper limit of normal (ULN)
    * Bilirubin >1.5 × ULN unless the participant has documented Gilbert syndrome (isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%)
    * Estimated glomerular filtration rate <60 mL/min/1.73 m2 (Modification of Diet in Renal Disease [MDRD])
15. QT interval corrected for heart rate using Fridericia's method (QTcF) > 450 msec at screening.
16. Contraindications to lumbar puncture including but not limited to lumbar scoliosis, coagulopathy, infection at site of puncture, use of anticoagulants at the time of study enrolment.
17. Participant with seizure disorder or history of seizures within 6 months.
18. Surgery within last 3 months or planned major surgery within next 3 months from the date of screening (other than minor cosmetic surgery and minor dental surgery).
19. Use or intended use of any medications/products known to alter drug absorption, metabolism, or elimination processes including St John's Wort within 4 weeks prior to receiving study drug and up to end of study. Use of such medication will be considered on a case-by-case basis as per the opinion of the Investigator and/or independent medical monitor.
20. Use of grapefruit or similar substances (Seville oranges or marmalade, grapefruit juice, grapefruit hybrids, pomelos, exotic citrus fruits or fruit juices) within 7 days prior to first dose of study drug until last dose administration.
21. Donation of blood or blood products within 3 months prior to screening.
22. History of, or positive screening test for, hepatitis C infection (defined as positive for hepatitis C virus antibody), hepatitis B infection (defined as positive for hepatitis B surface antigen), or human immunodeficiency virus I or II.
23. Use or intended use of any over-the-counter (vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) or prescription medications within 7 days or 5 half-lives (whichever is longer) prior to receiving study drug, with the exception of hormone replacement therapy and therapies for chronic stable diseases that have been stable for at least 30 days prior to screening and until Day 1, unless deemed acceptable by the Investigator.
24. Inability to be venipunctured or tolerate venous puncture.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the ALSFRS-R total score | From baseline to Week 12

SECONDARY OUTCOMES:
Time from baseline to the occurrence of either death, or permanent assisted ventilation | Baseline to Week 12 (>22 hours daily for >7 consecutive days), whichever comes first )
Change from baseline in slow vital capacity (SVC) | Baseline to Week 12
Change from baseline in serum neurofilament light chain biomarker | Baseline to Week 12
Number of patients with treatment emergent adverse events | Baseline to Week 12
Number of patients with Serious adverse event (SAE) | Baseline to Week 12
Cmax | baseline to Week 12
AUC | baseline to Week 12
Tmax | baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Deven Parmar, MD,FCP, Study Chair — Zydus Therapeutics Inc.
Locations (7):
- India (7):
  - Zydus Hospitals & Healthcare Research, Ahmedabad, Gujarat
  - Rhythm heart institute, Vadodara, Gujarat
  - BrainS Super Speciality Hospital, Bengaluru, Karnataka
  - KIMS-Kingsway Hospitals, Nagpur, Maharashtra
  - Surya Multispecialty Hospital, Nashik, Maharashtra
  - CIMET's Inamdar Multispeciality Hospital, Pune, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi

IPD SHARING:
Plan to Share IPD: No